CLINICAL TRIAL: NCT06262854
Title: Efficacy and Safety of aBIo- Absorbable Antibiotic Delivery in Calcium Sulphate Granules (Stimulan®) for the Treatment of Osteomyelitis in Patients With Diabetic FOOT: a Randomised, Double Blind, Controlled Clinical Study. The BIG D-FOOT Study
Brief Title: Efficacy and Safety of Stimulan® for the Treatment of Diabetic Foot Osteomyelitis. The BIG D-FOOT Study
Acronym: BIG D-FOOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Matteo Monami, MD, PhD, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOU Careggi Firenze
Record Dates: First submitted 2024-01-30; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Diabete Mellitus; Foot Ulcer; Osteomyelitis - Foot; Surgical Procedure, Unspecified
Keywords: diabetes;; foot osteomyelitis;; ulcer;; calcium sulphate local antibiotic delivery;; Stimulan
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Granules of calcium sulphate with and without antibiotics are identical and undistinguishable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Calcium-sulphate granules with tobramicina+vancomicina (Experimental)
  Interventions: Device: Calcium-sulphate granules with tobramicina+vancomicina
- Calcium-sulphate granules without antibioitcs (Sham Comparator)
  Interventions: Device: Calcium-sulphate granules with tobramicina+vancomicina

INTERVENTIONS:
Device: Calcium-sulphate granules with tobramicina+vancomicina — Local calcium-sulphate antibiotics deliver for the treatment of diabetic foot osteomyelitis

SUMMARY:
This study is designed as a double-blind, placebo-controlled, parallel series randomized trial aimed at verifying the effiicacy and safety of a local calcium-sulphate bio-absorbable antibiotic delivery (tobramicina+vancomicina) versus placebo (calcium-sulphate matrix without antibiotics) in patients with diabetic foot osteomyelitis treated with surgical procedures.

DETAILED DESCRIPTION:
Osteomyelitis is a severe complication of diabetic foot ulcers, that can occur in nearly 20-60% of patients. Current treatments for diabetic foot osteomyelitis (DFO) include surgical procedures aimed at removing necrotic soft tissue, gengrene and infected bones and systemic antibiotic therapy for at least 4-6 weeks; however in some cases, prolonged antibiotic therapy is not unusual.

Antibiotic therapy can be problematic for several reasons, such as the achievement of appropriate and stable therapeutic concentration at bone level, particularly due to the common presence of concomitant peripheral artery disease, and kidney impairment. In recent years, another important barrier to the treatment of DFO was the increasing incidence of resistant pathogens. On the other hand, surgical options are affected by several side effects, such as alterations of foot biomechanics possibly leading to new ulcers (the so called transfer ulcer), post-surgical infections, ecc. All these factors make the DFO treatment challenging, with a high risk of all-cause mortality and rate of patients requiring major amputations Local bio-absorbable antibiotic delivery can be a valid therapeutic option for DFO treatment. During the last 2 decades, biodegradable carriers have been developed: proteins (collagen, gelatin, thrombin etc.), synthetic polymers, grafts, and substitutes (calcium sulfate or phosphate).

Local antibiotic delivery system has been widely explored to increase the duration of local antibiotic delivery and bone penetration, achieving very high local therapeutical doses (about several times higher than that obtained with systemic antibiotic therapy) with reduced systemic toxicity. Another important advantage of this device is the possibility of using very effective, but highly toxic, antibiotic such as aminoglycosides, often not taken into account for systemic therapies.

Finally, this device can be used as a bone substitute filling the dead space caused by bone resection, thus reducing the incidence of reinfection. Complications of calcium sulfate are negligible and include postoperative drainage and transient hypercalcemia.

There several observational studies and very few randomized trials performed on DFO exploring the efficacy of local bio-absorbable antibiotic delivery and none on Stimulan.

The present study is designed as a double-blind, placebo-controlled, parallel series randomized trial aimed at verifying the effiicacy and safety of a local calcium-sulphate bio-absorbable antibiotic delivery (either with tobramicina or vancomicina) versus placebo (calcium-sulphate matrix without antibiotics) in patients with DFO treated with surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes
* Forefoot osteomyelitis
* Deep tissue infection

Exclusion Criteria:

* Pregnancy
* Severe cognitive impairment
* Creatinine clearance< 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The composite primary endpoint of this study will be the incidence osteomyelitis recurrence or new osteomyelitis in adjacent sites or tissue infection at the site of osteomyelitis. | 3 months
  Post-surgical infective complications

SECONDARY OUTCOMES:
Proportion of healed patients | 3 months
  Complete rehepitelization of the ulcer
Proportion of osteomyelitis recurrence | 3 months
  Recurrence of osteomyelitis in the same foot site
Proportion of post-surgical tissue infection | 3 months
  Tissue infection at the surgical wound level
Proportion of wound recurrence | 3 months
  New ulcer at the same site
Proportion of patients undergoing major amputation | 3 months
  Above ankle amputation
Proportion of patients undergoing new surgical intervention | 3 months
  New surgical intervention for osteomyelitis
Ulcer time-to-healing | 3 months
  From baseline to healing (days)
Osteomyelitis time-to-recurrence | 3 months
  From baseline to osteomyelitis recurrence (days)
Any serious adverse events | 3 months
  Life-threatening adverse events
Any non serious adverse events | 3 months
  Mild-moderate adverse events
Proportion of post-surgical dehiscence | 7 days
  Post-surgical infection
Direct medical costs | 3 months
  Costs for foot-related problems (hospital admission, amputation, revascularization, antibiotic therapy, medical device, etc.)